CLINICAL TRIAL: NCT01306968
Title: A Pilot Phase II Study of Hyperbaric Oxygen for Persistent Post-concussive Symptoms After Mild Traumatic Brain Injury (HOPPS)
Brief Title: Hyperbaric Oxygen Therapy (HBO2) for Persistent Post-concussive Symptoms After Mild Traumatic Brain Injury (mTBI)
Acronym: HOPPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S-10-09
Record Dates: First submitted 2011-02-24; First posted 2011-03-02 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Post-concussive Symptoms; Traumatic Brain Injury
Keywords: mild tramatic brain injury; mTBI; hyperbaric oxygen; post concussive symptoms; active duty military; veterans
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Injuries, Traumatic | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard TBI Care (No Intervention): Routine post-concussive symptoms (PCS) care as practiced within Departments of Defense (DoD)
- HBO2 Group (Experimental): Routine PCS care supplemented with hyperbaric oxygen (HBO2) at the dose of 1.5 ATA for 60 minutes administered over 40 sessions given daily Monday through Friday
  Interventions: Drug: hyperbaric oxygen
- Sham Group (Sham Comparator): Routine PCS care supplemented with an otherwise identical sham hyperbaric air exposure at 1.2 atmospheres absolute (ATA)
  Interventions: Other: sham hyperbaric air
- PTSD With no History of TBI (No Intervention): Subjects who have been diagnosed with PTSD but have no diagnosed or suspected brain injuries. This group does not receive HBO2.

INTERVENTIONS:
Drug: hyperbaric oxygen — The chamber will be compressed with air to 1.5 atm abs. Once the chamber is compressed to 1.5 atm abs, the subjects will don a hood and breathe 100% oxygen. Hoods will be supplied with oxygen with flows of at least 30 liters per minute and overboard dumping of excess gas. Each subject will complete 40 sessions.
  The duration of the hyperbaric oxygen exposures will be 60 minutes (±2 minutes), timed from when the chamber hatch or door closes, and ending when the chamber hatch or door opens ("door-to-door" time equals 60 minutes). The total intervention exposure time is 50 minutes (±2 minutes). The interval to compress to the intervention pressure (1.5 atm abs) and will be 5 minutes (±1 minute). The interval to decompress from the study pressure will be 5 minutes (±1 minute).
  Other Names: medical oxygen
  Arms: HBO2 Group
Other: sham hyperbaric air — A pressure of 1.2 atm abs will provide an equivalent inhaled oxygen concentration of 25%. The duration of the sham exposures will be 60 minutes (±2 minutes). Each subject will complete 40 sessions.
  Arms: Sham Group

SUMMARY:
This is a Phase II randomized trial designed to describe the magnitude of change between baseline and follow-up outcomes for symptom surveys and a battery of neuropsychological tests administered at time points corresponding before and after 10 weeks over observation in four groups:

* A military population with post-concussion syndrome (mTBI) receiving local standard care
* A military population with post-concussion syndrome (mTBI) receiving local standard care and sham hyperbaric oxygen sessions
* A military population with post-concussion syndrome (mTBI) receiving local standard care and hyperbaric oxygen at 1.5 atmospheres sessions
* A otherwise similar group with PTSD but no history of TBI receiving local standard care Differences and variability of the tests will be used for determining the optimum primary endpoint(s) for future trial, as well as for refinement of sample size and power calculations for these studies. The groups undergoing hyperbaric sessions will be assigned to receive HBO2 or sham using a randomized, double blind design.

Active duty military (Army, Marine, Navy, Air Force) men and non-pregnant women residing in the United States and who will remain in the military for the entire study period, aged 18-65 years who have been deployed one or more times to the US Central Command since the initiation of Operation Enduring Freedom (October 7, 2001) who either:

* have been diagnosed with Post Traumatic Stress Disorder (PTSD) as a result of traumatic events that occurred during the qualifying CENTCOM deployment, but have no diagnosed or suspected lifetime brain injuries resulting in loss or alteration of consciousness; OR
* have been diagnosed with at least one mild brain injury (mTBI) with persistent (> 4 months) symptoms sustained during one or more of those deployments

DETAILED DESCRIPTION:
Brain injury due to trauma is very common; nonetheless, no pharmacological therapy is known to improve outcomes. Medications are used to treat symptoms, such as seizures and affective disorders, but are not intended to affect the fundamental problem. If HBO2, which is regularly available and relatively safe, improves outcome in brain-injured subjects by treating the underlying pathophysiology of post-concussive syndrome, this would represent a significant advance in treatment of brain injury. Hyperbaric oxygen (HBO2) has been proposed as a treatment for patients with TBI.

Hyperbaric oxygen is one of the first pharmacologic interventions being tested in this population of individuals with mild TBI and chronic post-concussive symptoms targeted to improve cognition, memory, and functional status. However, much is unknown about how to measure improvement in post-concussive symptoms after an intervention in the targeted active duty population. In preparation for a pivotal efficacy study, the objectives of this study are to characterize two candidate primary outcome tools in our intended study population, the RPQ and the NSI, in order to better estimate the sample size needed to answer the efficacy question.

Agency for Healthcare Research and Quality (AHRQ) conducted a comprehensive review of the literature, interviewed subject matter experts (SME), and conducted focus groups with SMEs to evaluate the evidence for HBO2 for patients with TBI. The AHRQ concluded that "Although they are cited frequently, the case series and time-series studies of HBO2 for TBI patients had serious flaws. There were no high-quality studies of the use of HBO2 to improve function and quality of life in patients with chronic, stable disabilities from TBI. The most important gap in the evidence is a lack of a good quality time-series study or controlled trial of the effects of HBO2 on cognition, memory, and functional status in patients with deficits due to mild chronic TBI." Similarly, the Department of Health and Human Services (DHHS) has not approved HBO2 therapy for the treatment of TBI as a covered condition, citing the lack of supporting evidence for clinical efficacy.

The Defense Centers of Excellence for Psychological Health and Traumatic concluded that sufficient case reports, early safety and feasibility study data, and basic scientific plausibility exist to warrant prompt experimental study of HBO2 in the care of the full spectrum of chronic TBI. This would best be accomplished in a randomized, double-blind, multi-center clinical trial.

This Phase 2 study, through specific study design, inclusion and exclusion criteria, interim and end point analyses, treatment protocols, dose-response and safety issues, evaluation methodologies, safety, and outcome measures address the need for clinical efficacy.

In preparation for the pivotal trial, the purpose of this Phase II study is to describe the magnitude of change between baseline and follow-up outcomes for a battery of neuropsychological tests within groups. A secondary objective is to explore changes across the four groups. Differences and variability of the tests will be used for determining the optimum primary endpoint(s) for the Phase III trial, as well as for refinement of sample size and power calculations for this future study. Recruitment, randomization, blinding, and study and intervention logistics and planning will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have history of at least one mild traumatic brain injury (mTBI) with persistent symptoms that meets all the following criteria:

  * Brain injury that occurred more than 4 months prior to enrollment, with the most recent injury occurring no earlier than October 7, 2001.
  * Most recent traumatic brain injury occurred while serving on active duty, and while deployed to the United States (US) Central Command (USCENTCOM).
  * Most recent traumatic brain injury was caused by blast exposure or blunt trauma.
  * Most recent traumatic brain injury resulted in at least one of the following: a period of loss of or a decreased level of consciousness (up to 30 minutes); a loss of memory for events immediately before or after the injury (up to 24 hours); or alteration in mental state at the time of the injury (becoming dazed or confused).
* Volunteers must also meet all the following criteria:

  * 18-65 years old at the time of study enrollment.
  * A TRICARE beneficiary at the time of consent and during study participation.
  * Has current complaints of brain injury symptoms such as headache, dizziness, or cognitive or affective problems that score at least 3 post-concussive symptoms as assessed by the Ohio State University (OSU) Traumatic Brain Injury (TBI) Identification (ID) Method interview
  * Has received current local care pharmacologic and non-pharmacologic interventions for TBI and any concomitant posttraumatic stress disorder (PTSD) with no significant change in therapy for at least 1 month
  * Willing and committed to comply with the research protocol and complete all outcome measures.
  * Able to self-consent.
  * Able to speak and read English, as primary language.
  * Able to participate in all outcome measures.
  * Able to equalize middle ear pressure.

Exclusion Criteria:

* History of brain injury of moderate or severe degree: duration of loss of consciousness at the time of injury greater than 30 minutes, or duration of post-traumatic amnesia greater than 24 hours, or brain injury of a penetrating etiology.
* History of brain injury not of traumatic etiology, such as stroke or drug-induced coma.
* Prior treatment with HBO2.
* Hyperbaric chamber inside attendant, professional (paid)underwater diver (commercial, operational/ military, instructor), or technical diver.
* Pregnancy, women who plan to become pregnant during the study period, women who do not agree to practice an acceptable form of birth control during the study period, or women who are breastfeeding;
* Those who are unable to participate fully in outcome assessments (Blind in one or both eyes; Deaf in one or both ears; or Ambulation with assistive devices
* Pre-existing diagnosis of a psychotic disorder(s): schizophrenia, dissociative disorder, and bipolar disease.
* Verifiable degenerative mental disease (e.g., Alzheimer's disease, multiple sclerosis, senile dementia).
* Epilepsy or seizure disorder requiring anticonvulsants.
* Active malignancy, prior malignancy (except basal cell carcinoma) within the last 5 years.
* Presence of chronic debilitating disease (e.g., end-stage renal disease, end-stage liver disease, all types of diabetes with or without sequelae).
* Documented clinically significant uncorrected anemia
* Documented sickle cell disease.
* History of therapeutic ionizing radiation to the head.
* Verifiable diagnosis of learning disability.
* Positive urine test for an illicit substance(s).
* Any condition or use of prescribed medication (lithium, cisplatin, doxorubicin, or bleomycin) in which receipt of HBO2 would impact the safety of the individual.
* Anticipated administrative separation, prolonged temporary assigned duty (TAD/TDY) or deployment within 3 months after randomization
* Claustrophobia (unwilling or unable to enter hyperbaric chamber).
* Inability to protect airway or requires frequent suctioning; presence of tracheostomy
* Heart failure with ejection fraction < 50% (due to increased risk for precipitating acute lung edema during exposure to HBO2).
* Emphysema, chronic bronchitis, or bullous lung disease (due to risk for pulmonary barotrauma during hyperbaric decompression).
* Diabetes (relative contraindication related to risk of hypoglycemia).
* Presence of implanted device (e.g., cardiac defibrillator, intrathecal drug delivery device, cochlear implant) that poses increased risk to subject during hyperbaric exposure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Miller, MD, COL, Principal Investigator — United States Army Medical Materiel Development Activity
Locations (5):
- United States (5):
  - Naval Hospital Camp Pendleton, Camp Pendleton, California
  - Evans Army community Hospital Fort Carson, Fort Carson, Colorado
  - Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Naval Hospital Camp Lejeune, Marine Corps Base Camp Lejeune, North Carolina
  - Study Coordinating Center, LDS Hospital, Salt Lake City, Utah

REFERENCES:
- [Derived] Weaver LK, Churchill S, Wilson SH, Hebert D, Deru K, Lindblad AS. A composite outcome for mild traumatic brain injury in trials of hyperbaric oxygen. Undersea Hyperb Med. 2019 BIMA Special Edition No. Feb;46(3):341-352. PMID 31394603
- [Derived] Churchill S, Deru K, Weaver LK, Wilson SH, Hebert D, Miller RS, Lindblad AS. Adverse events and blinding in two randomized trials of hyperbaric oxygen for persistent post-concussive symptoms. Undersea Hyperb Med. 2019 BIMA Special Edition No. Feb;46(3):331-340. PMID 31394602
- [Derived] Miller RS, Weaver LK, Bahraini N, Churchill S, Price RC, Skiba V, Caviness J, Mooney S, Hetzell B, Liu J, Deru K, Ricciardi R, Fracisco S, Close NC, Surrett GW, Bartos C, Ryan M, Brenner LA; HOPPS Trial Team. Effects of hyperbaric oxygen on symptoms and quality of life among service members with persistent postconcussion symptoms: a randomized clinical trial. JAMA Intern Med. 2015 Jan;175(1):43-52. doi: 10.1001/jamainternmed.2014.5479. PMID 25401463

RESULTS

PARTICIPANT FLOW:
Groups:
- PTSD With no History of TBI: Non-randomized - Subjects who have been diagnosed with PTSD but have no diagnosed or suspected brain injuries. This group did not receive hyperbaric oxygen.
- HBO2 Group: Routine PCS care supplemented with hyperbaric oxygen (HBO2) at the dose of 1.5 ATA for 60 minutes administered over 40 sessions given daily Monday through Friday
  hyperbaric oxygen: The chamber will be compressed with air to 1.5 atm abs. Once the chamber is compressed to 1.5 atm abs, the subjects will don a hood and breathe 100% oxygen. Hoods will be supplied with oxygen with flows of at least 30 liters per minute and overboard dumping of excess gas. Each subject will complete 40 sessions.
  The duration of the hyperbaric oxygen exposures will be 60 minutes (±2 minutes), timed from when the chamber hatch or door closes, and ending when the chamber hatch or door opens ("door-to-door" time equals 60 minutes). The total intervention exposure time is 50 minutes (±2 minutes). The interval to compress to the intervention pressure (1.5 atm abs) and will be 5 minutes (±1 minute). The interval to decompress from the study pressure will be 5 minutes (±1 minute).
Period: Overall Study
Arm/Group | PTSD With no History of TBI | Standard TBI Care | HBO2 Group | Sham Group
Started | 7 | 23 | 24 | 25 (2 participants withdrew before chamber sessions were initiated)
Completed | 6 | 20 | 23 | 21
Not Completed | 1 | 3 | 1 | 4
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Relocated and left active duty | 0 | 1 | 1 | 1
Not completed — Withdrew - time commitment | 0 | 0 | 0 | 2
Not completed — Withdrew over privacy concerns | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTSD With no History of TBI | Standard TBI Care | HBO2 Group | Sham Group | Total
Number analyzed (Participants) | 7 | 23 | 24 | 25 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (9.0) | 30.3 (7.2) | 32.5 (7.9) | 31.4 (7.6) | 31.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 4
  Male | 6 | 22 | 23 | 24 | 75
Post-concussion Symptom Scores [Mean (Standard Deviation); unit: units on a scale] — The Rivermead Post-Concussion Symptom Questionnaire (RPQ) was created to measure the severity of post-concussion symptoms following traumatic brain injury (TBI). RPQ-3 are the first 3 symptoms of the RPQ Total including headaches, dizziness, and nausea/vomiting. RPQ-13 are the remaining 13 TBI symptoms. Using values of 0 (not experienced at all), 1 (no more of a problem than before the injury), 2 (mild problem), 3 (moderate problem), or 4 (severe problem). The range is 0 to 64. The score is a summation of symptoms rated as >2 representing new symptom onset or exacerbation of symptom(s).
  units on a scale
    RPQ-3 | 2.7 (1.89) | 5.4 (2.74) | 5.5 (3.27) | 4.7 (3.09) | 5.0 (3.01)
    RPQ-13 | 20.9 (9.19) | 27.1 (12.20) | 27.5 (13.15) | 25.5 (11.61) | 26.2 (12.02)
    RPQ Total | 23.6 (10.11) | 32.5 (14.39) | 33.0 (15.82) | 30.2 (14.17) | 31.1 (14.55)

OUTCOME MEASURES:

1. Primary Outcome: Post-Intervation Post-concussion Symptom Scores Using RPQ - Intent to Treat
Description: The Rivermead Post-Concussion Symptom Questionnaire (RPQ)/RPQ-3 was created to measure the severity of post-concussion symptoms following traumatic brain injury. The scale compares any current symptoms to pre-injury levels to account for potential symptom exacerbation due to the TBI. The RPQ is the most commonly used clinical outcome measure for mild TBI research because it is simple and reflects psychosocial function. The RPQ is intended to measure the presence and severity of 16 of the most commonly reported post-concussion symptoms found in the literature.
Time Frame: Follow-up Visit 2; Day 56 (up to day 100) for groups not recieving HBO2, Day 70 for groups recieving HBO2
Population: Intent to treat population: All randomized participants were included in the intention-to-treat analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- HBO2 Group: Routine PCS care supplemented with hyperbaric oxygen (HBO2) at the dose of 1.5 ATA for 60 minutes administered over 40 sessions given daily Monday through Friday. Each subject will complete 40 sessions.
  The duration of the hyperbaric oxygen exposures will be 60 minutes (±2 minutes), timed from when the chamber hatch or door closes, and ending when the chamber hatch or door opens ("door-to-door" time equals 60 minutes). The total intervention exposure time is 50 minutes (±2 minutes). The interval to compress to the intervention pressure (1.5 atm abs) and will be 5 minutes (±1 minute). The interval to decompress from the study pressure will be 5 minutes (±1 minute).
Arm/Group | PTSD With no History of TBI | Standard TBI Care | HBO2 Group | Sham Group
Number analyzed (Participants) | 6 | 20 | 23 | 21
units on a scale
  RPQ-3 | 3.5 (3.21) | 5.1 (2.81) | 4.2 (3.00) | 3.5 (3.25)
  RPQ-13 | 19.7 (13.06) | 25.5 (13.93) | 22.5 (12.35) | 20.7 (12.82)
  Total RPQ | 23.2 (16.04) | 30.6 (16.08) | 26.7 (24.83) | 24.2 (15.38)

2. Primary Outcome: Change in Post-concussion Symptom Scores Using RPQ - Intent to Treat
Description: Means for the change from baseline to follow-up visit 2
Time Frame: Follow-up Visit 2; Day 56 (up to day 100) for groups not recieving HBO2, Day 70 for groups recieving HBO2
Population: Intent to treat population: All randomized participants were included in the intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard TBI Care: Routine post-concussive symptoms (PCS) care as practiced within Departments of Defense (DoD) Follow-up visit 2 = Day 56 (up to day 100)
Arm/Group | PTSD With no History of TBI | Standard TBI Care | HBO2 Group | Sham Group
Number analyzed (Participants) | 6 | 20 | 23 | 21
units on a scale
  RPQ-3 | 0.3 (2.73) | 0.0 (2.05) [-0.96 to 0.96] | -1.2 (2.81) [0.0 to 2.43] | -1.5 (3.01) [0.11 to 2.85]
  RPQ-13 | -3.0 (15.39) | -0.5 (9.65) [-4.0 to 5.0] | -4.2 (11.42) [-0.8 to 9.1] | -5.5 (10.50) [0.7 to 10.3]
  Total RPQ | -2.7 (17.88) | -0.5 (11.32) [-4.8 to 5.8] | -5.4 (13.66) [-0.5 to 11.3] | -7.0 (12.97) [1.0 to 12.9]

3. Primary Outcome: Post-Intervation Post-concussion Symptom Scores Using RPQ - Per Protocol Population
Description: as for outcome 1
Time Frame: Follow-up Visit 2; Day 56 (up to day 100) for groups not recieving HBO2, Day 70 for groups recieving HBO2
Population: Per protocol population: Only those completing all 40 chamber sessions and outcomes testing are included in the per protocol population. The standard TBI care group remained the same as no champber sessions were use in this group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTSD With no History of TBI | Standard TBI Care | HBO2 Group | Sham Group
Number analyzed (Participants) | 6 | 20 | 11 | 13
units on a scale
  RPQ-3 | 3.5 (3.21) | 5.1 (2.81) | 3.1 (2.21) | 2.7 (2.84)
  RPQ-13 | 19.7 (13.06) | 25.5 (13.93) | 15.6 (10.93) | 17.4 (13.25)
  Total RPQ | 23.2 (16.04) | 30.6 (16.08) | 18.7 (12.96) | 20.1 (15.67)

4. Primary Outcome: Change in Post-concussion Symptom Scores Using RPQ - Per Protocol Population
Description: as for outcome 1
Time Frame: Follow-up Visit 2; Day 56 (up to day 100) for groups not recieving HBO2, Day 70 for groups recieving HBO2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PTSD With no History of TBI | Standard TBI Care | HBO2 Group | Sham Group
Number analyzed (Participants) | 6 | 20 | 11 | 13
units on a scale
  RPQ-3 | 0.3 (2.73) | 0.0 (2.05) [lower limit 2.05] | -1.6 (2.54) | -2.2 (2.44)
  RPQ-13 | -3.0 (15.39) | -0.5 (9.65) [-4.0 to 5.0] | -9.4 (9.68) [2.9 to 15.9] | -8.5 (9.44) [2.8 to 14.2]
  Total RPQ | -2.7 (17.88) | -0.5 (11.32) [-4.8 to 5.8] | -11.0 (11.64) [3.2 to 18.8] | -10.7 (11.22) [3.9 to 17.5]

ADVERSE EVENTS:
Time Frame: Within 14 days of the last chamber session
Description: Standard TBI Care and PTSD with no history of TBI groups recieved no HBO2 exposure and were not at risk for chamber intervention related injury. 2 participants withdrew before chamber sessions were initiated. Safety population of HBO2 (n=24) and sham (n=23)
Arm/Group | PTSD With no History of TBI | Standard TBI Care | HBO2 Group | Sham Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 8/24 | 6/23
OTHER ADVERSE EVENTS (reported when occurring in more than 4.2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTSD With no History of TBI (N=0) | Standard TBI Care (N=0) | HBO2 Group (N=24) | Sham Group (N=23)
mild ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inner ear barotrauma (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Onset migraine headache (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increase frequency and intensity of headaches (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient worsening of myopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Change in headache frequency (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Claustrophobia/anxiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No